CLINICAL TRIAL: NCT06157294
Title: Comparison of the Treatment Outcomes of the Facet Intra-articular Pulsed Radiofrequency and Median Branch Pulsed Radiofrequency Interventions in Lumbar Facet-related Pain
Brief Title: Pulsed Radiofrequency Treatment in Lumbar Facet-Related Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Başakşehir Çam & Sakura City Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2021.05.102
Record Dates: First submitted 2023-11-27; First posted 2023-12-05 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-11

CONDITIONS: Facet Joint Pain; Pain Syndrome; Pain, Chronic
MeSH Terms: conditions — Somatoform Disorders; Chronic Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intra-articular pulsed radiofrequency group (Active Comparator): This arm consists of patients who received intra-articular pulse radiofrequency treatment.
  Interventions: Procedure: Intra-articular pulsed radiofrequency
- Median branch pulsed radiofrequency group (Active Comparator): This arm consists of patients who received median branch pulse radiofrequency treatment.
  Interventions: Procedure: Median branch pulsed radiofrequency

INTERVENTIONS:
Procedure: Intra-articular pulsed radiofrequency — Intra-articular pulsed radiofrequency procedures for the treatment of facet joint-related low back pain are performed under sterile conditions in the operating room. The application is performed under fluoroscopy guidance using a 20 gauge 10 mm active tip radiofrequency needle. When the intra-articular joint, which is the target tissue, is reached with the help of fluoroscopy images, pulse radiofrequency treatment will be applied with the parameters being maximum temperature 42 degrees, 45 volts, duration 6 minutes, pulse rate 2 hertz and pulse width 20 milliseconds.
  Arms: Intra-articular pulsed radiofrequency group
Procedure: Median branch pulsed radiofrequency — Median branch pulsed radiofrequency procedures for the treatment of facet joint-related low back pain are performed under sterile conditions in the operating room. The application is performed under fluoroscopy guidance using a 20 gauge 10 mm active tip radiofrequency needle. When the median branch region, which is the target area, is reached with the help of fluoroscopy images, location confirmation will be provided by giving sensory and motor stimulation. Pulse radiofrequency treatment will be applied with the parameters being maximum temperature 42 degrees, 45 volts, duration 6 minutes, pulse rate 2 hertz and pulse width 20 milliseconds.
  Arms: Median branch pulsed radiofrequency group

SUMMARY:
Facet joint-related pain is one of the leading causes of low back pain. Facet joint-related disorders can have a negative impact on quality of life and daily living activities, in addition to the pain.Conservative treatment methods such as analgesic medications, physical therapy, and manual therapy are used for facet joint-related low back pain, and interventional pain management practices are used in patients who do not respond adequately to these treatments.

Pulse radiofrequency application, which is a recent popular treatment in interventional pain management, is also frequently applied in the treatment of facet-joint related pain. Pulsed radiofrequency intervention can be applied directly intra-articularly or can be applied to the median branch, which is important structure in pain transmission. Although both methods are frequently used in pain management, there is a lack of information in the literature about which is more effective. This study aimed to compare the treatment results of intraarticular pulse radiofrequency application and median branch pulse radiofrequency application in facet joint-related low back pain.

ELIGIBILITY:
Inclusion Criteria:

* Having facet joint-related low back pain at least 3 months
* No response to other conservative treatments (analgesic medications, physical therapy, manuel therapy etc.)
* Patients with a pain severity score of at least 6 according to NRS

Exclusion Criteria:

* History of lumbar region surgery
* Patients with bleeding disorders
* Presence of pregnancy and breastfeeding status
* Presence of the infection related findings and any other systemic disorder
* History of allergic reaction to contrast agent
* Patients who do not have sufficient mental function to fill out the scales during the follow-up periods

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-11-27 (Actual)

PRIMARY OUTCOMES:
Change of the pain severity score | Pre-intervention, post-intervention 1th month and post-intervention 6th month
  Pain severity is assessed by using "Numeric Rating Scale" (NRS). Patients give score of their pain between 0 (no pain) and 10 (worst possible pain). The change in NRS scores between the two groups will be compared.

SECONDARY OUTCOMES:
Change of the disability score | Pre-intervention, post-intervention 1th month and post-intervention 6th month
  Disability conditions of the patients are assessed by using "Oswestry Disability Index" (ODI). ODI is a patient-completed questionnaire which gives a percentage score of disability. The ODI is comprised of 10 items and enquires about functional limitations in various activities of daily living with the index score ranging from 1 (best) to 100 (worst). The change in ODI scores between the two groups will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Burak Erken, MD, Principal Investigator — Başakşehir Çam & Sakura City Hospital
Locations (1):
- Basahsehir Cam and Sakura City Hospital, Istanbul, Turkey (Türkiye)